CLINICAL TRIAL: NCT01224990
Title: Whole Body Diffusion MRI for Non-invasive Lesion Detection and Therapy Follow-up: Study With Patients With Gastro-intestinal Tumors.
Acronym: s51240
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, katrijn Michielsen, PhD department of Radiology, Universitaire Ziekenhuizen KU Leuven
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: s51240
Record Dates: First submitted 2010-10-19; First posted 2010-10-20 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: Gastro-intestinal Tumor; Accurate Staging; Whole-body Diffusion Weighted MRI; Non-invasive
Keywords: gastro-intestinal tumor; accurate staging; whole-body diffusion weighted MRI; non-invasive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Whole body diffusion MRI — These studies will be performed on a 3Tesla (T) MR system (Achieva, Philips Medical Systems). A major advantage of 3T compared to 1.5 T is the improved signal to noise ratio that allows whole-body studies to be faster and without application of external antennas, which greatly improves patient comfort.

SUMMARY:
The aim of the study is to assess the value of whole body diffusion weighted MR imaging (WB-DWI) as a non-invasive method. On one hand for pretreatment lesion detection and post-therapeutic tumor recurrence but also for early therapy monitoring with the intention to early identify patients with a poor tumor response. Our research group demonstrated that this technique is accurate in patients with head and neck cancer it could differentiate between viable tumor tissue and inflammatory or necrotic tissue at variable time points after completion of radiotherapy. In the literature it is stated that DWI can also predict the response to chemotherapeutic therapy. This is only true for focal MRI images (eg only in liver). This study aims to determine whether the whole body technique can efficiently be used because the distribution of metastases is systemic. The study includes two phases: In a first phase, a baseline study will be conducted; all possible injury types will be gathered to determine the variability in signal characteristics to finally determine appropriate thresholds to differentiate between benign and malignant lesions. This should allow us later on to perform prospective studies. In a second phase, different applications such as:

* pretherapeutic staging
* Detection of post-therapy recurrence
* Early evaluation of systemic cytotoxic therapy.

The results of the DW-MRI will be compared with those of PET, CT and conventional MRI which are now routinely performed for the diagnosis of colorectal tumors. The scans will be performed in a group of patients on a 3 Tesla MR system. This system is fully approved by the European and American standards and the patients will not be exposed to radiation or contrast agents. In principle, all patients treated for gastrointestinal cancer were included after informed consent from the patient. This study is important to investigate whether DWI is accurate in the pre-therapeutic injury detection and staging of gastrointestinal tumors compared with PET / CT and DWI. In addition it is important to predict the outcome after therapy.

ELIGIBILITY:
Inclusion Criteria:

* In principle, all patients treated for gastrointestinal tumors will be included (only with the permission (informed consent) of the patient)

Exclusion Criteria:

* In case of a known contraindication for MRI (eg pacemaker), the patient will not be admitted to the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2010-11; Primary Completion 2014-11 (Actual); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
The aim of the study is to asses whole body diffusion weighted imaging (WB-DWI) in patients with proven gastro-intestinal tumors and to evaluate this non-invasive method for staging and therapy monitoring. | The outcome measure will be assessed during the whole study period (2010-2014)
  The aim of the study is to asses whole body diffusion weighted imaging (WB-DWI) in patients with proven gastro-intestinal tumors and to evaluate this non-invasive method for staging and therapy monitoring.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Gasthuisberg, Leuven, Leuven, Belgium